CLINICAL TRIAL: NCT04710563
Title: SCOPE-CLI: Shifting Care and Outcomes for Patients With Endangered Limbs - Critical Limb Ischemia
Brief Title: SCOPE-CLI: Shifting Care and Outcomes for Patients With Endangered Limbs
Acronym: SCOPE-CLI
Status: Active, not recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: University of Chicago (Other); Oregon Health and Science University (Other); University of California, Davis (Other); University of Southern California (Other); Baylor College of Medicine (Other); The Cleveland Clinic (Other); Emory University (Other); Brown University (Other); Columbia University (Other); University of Minnesota (Other); Saint Luke's Health System (Other); Abbott (Industry); Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2000028963; 000 (Other: CTGTY)
Record Dates: First submitted 2021-01-04; First posted 2021-01-14 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A research project capturing experiences of patients with critical limb threatening ischemia, with the ultimate goal of setting new standards for diagnosing, describing detailed patient-centered outcomes, and evaluating the variability in therapeutic approaches and their association with outcomes.

DETAILED DESCRIPTION:
An estimated 8 million individuals in America are affected by peripheral arterial disease (PAD). One of its extreme expressions is Critical Limb Ischemia (CLI). It is one of the most severe vascular conditions associated with devastating outcomes, including poorly healing wounds, extreme pain, and a high amputation risk. It is also one of the deadliest conditions, with 6-month and 5-year mortality rates estimated to be 20 and >50%, respectively. To date, however, there is a paucity of prospective clinical evidence about the variability in patients' presentations, their management or their outcomes. Accordingly, little progress has been made in adequately staging the disease and to risk-stratify treatment approaches to patients' individual characteristics. What is desperately needed to advance the care and management of patients with CLI is a focused research effort to set new standards for diagnosing, describing detailed patient-centered outcomes, and evaluating the variability in therapeutic approaches and their association with outcomes. The specific aims of SCOPE-CLI are to generate new evidence on the clinical characteristics, treatment patterns and outcomes of patients with critical limb ischemia (CLI); to describe treatment patterns and variability across practices to identify gaps in delivering quality care; and to perform a series of analyses to examine the associations of patient and treatment characteristics with outcomes. The central objective of SCOPE-CLI is to systematically quantify patients' CLI-specific health status and clinical outcomes and to perform subgroup analyses as a function of different PAD treatments and patient characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. All race/ethnicity categories, English speaking, men and women
2. Patient presents with current (within 30 days) Rutherford Class 4, 5, or 6
3. Age ≥18 years
4. Supported by any of the following diagnostic evidence:

   * Rutherford Classification 4 or ischemic rest pain and/or resting ankle pressure <50mmHg, flat or barely pulsatile ankle or metatarsal PVR or toe pressure <40mmHg
   * Rutherford Classification 5 or minor tissue loss; non-healing ulcer, focal gangrene with diffuse pedal ischemia resting ankle pressure <50mmHg ankle or metatarsal PVR flat or barely pulsatile or toe pressure <40mmHg
   * Rutherford Classification 6 or major tissue loss: extending above transmetatarsal level, functional foot no longer salvageable, resting ankle pressure <50mmHg ankle or metatarsal PVR flat or barely pulsatile or toe pressure <40mmHg
   * CLI related ICD 10 code (reason for admission or indication for procedure)
   * SPP < 50 mmHg
   * TCPO2 < 50 mmHg
   * Angiographic evidence no straight line to foot or greater than 70% stenosis in all 3 lower extremity arteries (AT, PT, peroneal)
   * ABI* ≤ 0.90
   * non-compressible ABI ≥ 1.40 AND TBI ≤ 0.70
   * TBI* ≤ 0.70

Exclusion Criteria:

1. Acute limb ischemia
2. Unable to provide written informed consent
3. Currently a prisoner (identified at time of enrollment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled from a range of clinical practices combining forces from vascular surgery, vascular medicine (interventional) cardiology, wound care specialists and podiatry clinics that treat CLI patients. All patients will be medically stable, i.e., not actively experiencing a life-threatening critical condition for which emergent care processes are ongoing, before they are approached for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Peripheral Artery Questionnaire (PAQ) | After enrollment and follow-up at month 1
  PAD-specific, multi-dimensional health status instrument with a CLI specific module. Higher scores indicate better functioning.
Peripheral Artery Questionnaire (PAQ) | After enrollment and follow-up at month 2
  PAD-specific, multi-dimensional health status instrument with a CLI specific module. Higher scores indicate better functioning.
Peripheral Artery Questionnaire (PAQ) | After enrollment and follow-up at month 6
  PAD-specific, multi-dimensional health status instrument with a CLI specific module. Higher scores indicate better functioning.
Peripheral Artery Questionnaire (PAQ) | After enrollment and follow-up at month 12
  PAD-specific, multi-dimensional health status instrument with a CLI specific module. Higher scores indicate better functioning.

SECONDARY OUTCOMES:
Major adverse limb events (MALE) | 6 months after enrollment
  Major adverse limb events include: major amputation above the level of the ankle joint, thrombolysis/thrombectomy or surgical bypass or graft revision, after diagnostic or interventional lower extremity angiography)
Major adverse limb events (MALE) | 12 months after enrollment
  Major adverse limb events include: major amputation above the level of the ankle joint, thrombolysis/thrombectomy or surgical bypass or graft revision, after diagnostic or interventional lower extremity angiography)
Major adverse limb events (MALE) | 5 years after enrollment
  Major adverse limb events include: major amputation above the level of the ankle joint, thrombolysis/thrombectomy or surgical bypass or graft revision, after diagnostic or interventional lower extremity angiography)
Amputation Free Survival (AFS) | 6 months after enrollment
  AFS will be a measure of number of patients "free from death or above ankle amputation"
Amputation Free Survival (AFS) | 12 months after enrollment
  AFS will be a measure of number of patients "free from death or above ankle amputation"
Amputation Free Survival (AFS) | 5 years after enrollment
  AFS will be a measure of number of patients "free from death or above ankle amputation"
Mortality - Death | 6 months after enrollment
  Vital status obtained from either medical records or social security death index will be assessed to account for number of patients who died
Mortality - Death | 12 months after enrollment
  Vital status obtained from either medical records or social security death index will be assessed to account for number of patients who died
Mortality - Death | 5 years after enrollment
  Vital status obtained from either medical records or social security death index will be assessed to account for number of patients who died

CONTACTS AND LOCATIONS:
Overall Officials: Kim Smolderen, PhD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Health, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Scierka LE, Mena-Hurtado C, Shishehbor MH, Spertus JA, Nagpal S, Babrowski T, Bunte MC, Politano A, Humphries M, Chung J, Kirksey L, Alabi O, Soukas P, Parikh S, Faizer R, Fitridge R, Provance J, Romain G, McMillan N, Stone N, Scott K, Fuss C, Pacheco CM, Gosch K, Harper-Brooks A, Smolderen KG; SCOPE-CLI Academic Research Consortium. The shifting care and outcomes for patients with endangered limbs - Critical limb ischemia (SCOPE-CLI) registry overview of study design and rationale. Int J Cardiol Heart Vasc. 2022 Feb 12;39:100971. doi: 10.1016/j.ijcha.2022.100971. eCollection 2022 Apr. PMID 35198727